CLINICAL TRIAL: NCT02124434
Title: Laparoscopic Sleeve Gastrectomy - A Prospective Study of Weight Loss, Comorbidities and Patients' Quality of Life
Status: Completed | Type: Observational
Sponsor: Meir Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: MMC14062-13CTIL
Record Dates: First submitted 2014-04-06; First posted 2014-04-28 (Estimated); Last update posted 2018-03-22 (Actual); Status verified 2018-03

CONDITIONS: Obesity
Keywords: Laparoscopic Sleeve Gastrectomy surgery
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Laparoscopic Sleeve Gastrectomy: Patients undergoing Laparoscopic Sleeve Gastrectomy surgery for morbid obesity

SUMMARY:
Surgery is considered the best therapy for morbid obesity and its comorbidities, where alterations in lifestyle, diets and drugs have failed to achieve weight loss. The most widely performed in Israel is Laparoscopic Sleeve Gastrectomy (LSG), and several studies have reported high success rates in reducing weight and improving comorbidities common among obese patients such as hypertension; diabetes mellitus type II; dyslipidemia; osteoarthritis; obstructive sleep apnea etc.

The hypothesis of this prospective study is that the LSG is an effective treatment for achieving weight loss, for improving and even curing comorbidities and for improving the patient's QOL. Another supposition is that patient's socio-economic status can influence success rates of bariatric procedures.

DETAILED DESCRIPTION:
Introduction - Morbid obesity is considered an ever growing pandemic. Most morbidly obese patients suffer from comorbidities such as hypertension; diabetes mellitus type II; dyslipidemia; osteoarthritis; obstructive sleep apnea etc. Surgery is considered the best therapy for morbid obesity and its comorbidities, where alterations in lifestyle, diets and drugs have failed to achieve weight loss. There are some procedures, some more commonly practiced than others, most of them done laparoscopically. The most widely performed in Israel is Laparoscopic Sleeve Gastrectomy (LSG), and several studies have reported high success rates in reducing weight and improving comorbidities. However, few studies exists, mostly retrospective, on the long term results after LSG. These studies have demonstrated significant weight loss, significant decrease in excessive body weight and also significant improvement in patients' quality of lives (QOL). However, a single comprehensive prospective research encompassing all three parameters was not found by us in a preliminary literature review. No studies were found regarding the effect of socio-economic status on the late results of LSG.

Goals -The goal of the present study is to prospectively follow patients undergoing LSG and to assess its effectiveness in weight loss and in the improvement of comorbidities and quality of life. We also plan to evaluate the effect of socio-economic status on the results of bariatric surgery, with emphasis on changes in QOL of these patients.

Material and Methods - In an 18 month long prospective research, a set of two questionnaires will be given to each patient undergoing LSG for morbid obesity at three time points: before surgery, 6 and 12 months post-surgery. The first questionnaire includes demographic, socio-economic and physiological data and health related questions regarding comorbidities and their methods of treatment. The second questionnaire is the Short Form 36v2, an accepted QOL questionnaire which, using 36 questions. At the end of the research, a statistical analysis of the results will be performed.

Hypothesis - The hypothesis states that the LSG is an effective treatment for achieving weight loss, for improving and even curing comorbidities and for improving the patient's QOL. Another supposition is that patient's socio-economic status can influence success rates of bariatric procedures.

Importance of the study - Several studies was done reviewing this procedure's efficacy according to physiological parameters and improvement in comorbidities and quality of life. Most of which are retrospective. A prospective research that encompasses all these three parameters was not currently found in the medical literature Keywords - Morbid Obesity, Bariatric surgery, Sleeve Gastrectomy, Quality of Life, Comorbidities, Weight loss.

ELIGIBILITY:
Inclusion Criteria:

* age between 18-70

Exclusion Criteria:

* patients who underwent previous bariatric surgery
* patients unwilling to participate in the study
* female patients who are currently pregnant
* patients who are cognitively impaired or lacking judgement

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing Laparoscopic Sleeve Gastrectomy surgery for morbid obesity.
Sampling Method: Non-Probability Sample
Enrollment: 97 (Actual)
Dates: Start 2014-02; Primary Completion 2015-10-30 (Actual); Study Completion 2015-10-30 (Actual)

PRIMARY OUTCOMES:
Weight loss | 1 year
  Observe and record subjects' weight loos over the course of one year.
Improvement in quality of life | 1 year
  observe and record the improvement in subjects' quality of life as reported by them in the questionnaire

SECONDARY OUTCOMES:
Improvement in comorbidities | 1 year
  Observe and record improvement in five obesity related comorbidities -
  * Diabetes mellitus type 2
  * Hypertension
  * Dyslipidemia
  * Osteoarthritis
  * Obstructive sleep apnea

OTHER OUTCOMES:
The affect of education, socioeconomic status and ethnic origin on the results of the surgery | 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Meir Medical Center, Kfar Saba, Israel